CLINICAL TRIAL: NCT00186407
Title: High Dose Chemotherapy and Autologous Stem Cell Rescue for Primary Amyloidosis
Brief Title: Autologous Stem Cell Rescue for Primary Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sally Arai, Stanford University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMT92; 76379; BMT92; NCT00186407
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Amyloidosis; Blood and Marrow Transplant (BMT)
MeSH Terms: conditions — Amyloidosis

INTERVENTIONS:
Procedure: high dose chemo then auto hematopoietic cell transplant

SUMMARY:
To evaluate the role of high dose therapy and autologous hematopoietic cell transplant for amyloidosis.

DETAILED DESCRIPTION:
To learn about the use of high dose chemotherapy followed by transplantation using peripheral blood stem cells.

ELIGIBILITY:
Inclusion Criteria:1. Primary amyloidosis

2. Age < 75 years.

3. Patients must have their pathology reviewed and the diagnosis confirmed at Stanford University Medical Center.

4. Patients who have undergone bone marrow transplantation previously will not be eligible.

5. Patients must have a Karnofsky performance status greater than 70%.

6. Patients must have a serum creatinine less than 2 mg/dl or creatinine clearance greater than 30 ml/min, bilirubin less than 2 mg/dl, transaminases less than two times normal, left ventricular ejection fraction >45% on echocardiography, cardiac index > 1.8 liters/min/m^2 and pulmonary function tests demonstrating FEV1 and DLCO > 60%.

7. Patients must be HIV negative.

8. Pregnant or lactating women will not be eligible to participate.

9. Patients must provide signed informed consent.

10. Patients with multiple myeloma and amyloid are eligible.

Exclusion Criteria:1. prior blood or marrow transplant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 1998-04; Primary Completion 2008-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the role of high dose therapy and autologous hematopoietic cell transplant for amyloidosis

CONTACTS AND LOCATIONS:
Overall Officials: Sally Arai, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States